CLINICAL TRIAL: NCT04097132
Title: Pattern of Non Valvular Atrial Fibrillation in Acute Ischemic Stroke Patients at Assiut University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shery Refaat Asaad, principal investigator, Assiut University
Other Study IDs: Pattern of non valvular AF
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Echocardiography; Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ischemic stroke patients: all patient admitted with acute ischemic stroke either their ECG was AF or sinus rythm
  Interventions: Device: echocardiography

INTERVENTIONS:
Device: echocardiography — echocardiography for left atrial diameter, size ,Ejection Fraction Holter for detection of paroxusmal AF
  Other Names: holter

SUMMARY:
Pattern of non valvular Atrial fibrillation in acute ischemic stroke patients at Assiut University Hospitals.

DETAILED DESCRIPTION:
Percentage of patients with AF admitted with acute cerebrovascular stroke at Assuit University and correlation between AF and severity of stroke at admission and discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with acute cerebrovascular stroke aged more than 18 years old.

Exclusion Criteria:

1. Patients below 18 years old.
2. Patient admitted with cerebral hemohrrage.
3. Patients with significant valvular heart disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all cases of acute cerebrovascular stroke in Assiut university hospital
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with AF admitted with acute cerebrovascular stroke at Assuit University. | 1 year
  study the Percentage of patients with AF admitted with acute cerebrovascular stroke at Assuit University whatever those patients have manifest atrial fibrillation or go into attacks of paroxysmal atrial fibrillation by the use of echocardiography for measurement of left atrial diameter and size and also by the use of Holter to identify any any attacks of paroxysmal atrial fibrillation

SECONDARY OUTCOMES:
correlation between AF and severity of stroke at admission and discharge. | 1 year
  relation between presence of AF and severity of stroke by the use of NIH Stroke Score and MRS score at time of admission and discharge.
The role of anti coagulants in decreasing risk of ischemic cerebrovascular stroke in patients who are known to have Atrial Fibrillation and have been already anticoagulated | 1 year
  if the anticoagulant intake decrease stroke severity in patients who are already taking anticoagulants by the use of NIH Stroke Score and MRS score at time of admission and discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Shery Refaat Asaad, Asyut, Egypt